CLINICAL TRIAL: NCT06500520
Title: Comparison of the Effects of Resistant Exercise and Stretching Exercises on Menstrual Symptoms, Quality of Life, Functional and Emotional Status in Young Women With Primary Dysmenorrhea
Brief Title: Resistive Exercise and Stretching in Women With Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: women Health
Record Dates: First submitted 2024-06-27; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Dysmenorrhea Primary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resisted Exercise group (Active Comparator): Participants underwent resistance training for 8 weeks, focusing on trunk, upper, and lower body segments with 10-12 reps per exercise at 30-65% intensity. Sessions lasted 50-60 minutes, 3 times weekly
  Interventions: Other: Resisted Exercise group
- Stretching Exercise group (Active Comparator): The participants were made to perform stretching exercises, selected by reviewing the literature, under supervision 3 days a week for 8 weeks, and they were asked not to do any other exercises during this intervention period.
  Interventions: Other: Stretching Exercise group
- control group (No Intervention): No treatment was applied to the control group; they were allowed to use painkillers and continued their normal daily lives.

INTERVENTIONS:
Other: Resisted Exercise group — The resisted exercise training program targeted trunk, upper, and lower body segments with 10-12 repetitions at 30-65% intensity, lasting 50-60 minutes per session, 3 times weekly for 8 weeks. Participants determined their maximal repetition through trial training. Maximal power was assessed using concentric 1-maximal repetition (MT). Following a 2-3 minute rest and a 5-minute warm-up (walking), participants performed the 1-MT test to establish their heaviest lift with the correct technique, adjusting resistance levels accordingly. The circuit-style training spanned 9 stations with 2-3 sets per station, each circuit lasting 2-3 minutes with 90-second rests between sets. A 5-minute warm-up and cool-down (walking) preceded and followed each session. Exercises included bilateral elbow flexion, chest press, bilateral shoulder abduction, bilateral knee extension, back extension, sit-ups, knee flexion, hip abduction, and hip adduction.
  Arms: Resisted Exercise group
Other: Stretching Exercise group — The participants were made to perform stretching exercises, selected by reviewing the literature, under supervision 3 days a week for 8 weeks, and they were asked not to do any other exercises during this intervention period. They were asked to do exercises such as trunk flexion, pelvic elevation, squatting, trunk lateral flexion, lumbar extensor stretching, lower abdominal stretching, hip adduct stretching, piriformis stretching, and trunk flexor stretching (cobra pose). The holding time was 5 seconds, the rest time was 1 second, and the exercises were applied in 10 repetitions.
  Arms: Stretching Exercise group

SUMMARY:
This study highlights the importance of exercise for young women with primary dysmenorrhea. Exercise can help relieve the symptoms of dysmenorrhea by increasing blood flow and promoting the release of endorphins. Additionally, exercise can improve the overall quality of life by reducing stress and anxiety. A comprehensive comparison of the effects of especially resistant exercises and stretching exercises on menstrual pain is based on limited findings in the literature. Therefore, this study aims to make a significant contribution to clinical practice by evaluating the effectiveness and feasibility of these exercise types.

DETAILED DESCRIPTION:
Primary dysmenorrhea is a common condition that seriously affects women's quality of life, and alternative methods other than pharmacotherapy are often investigated. Exercise may play a potential role in reducing the symptoms of dysmenorrhea by increasing blood flow and promoting the release of endorphins. Additionally, exercise can improve the overall quality of life by reducing stress and anxiety. However, studies comparing the specific effects of resistance exercises and stretching exercises on dysmenorrhea are limited and do not provide clear guidance on this subject. The aim of this study is to evaluate the effectiveness and feasibility of these two types of exercise in young women with primary dysmenorrhea. The results of the research can guide healthcare professionals by providing information on which type of exercise may be more effective in clinical practice. The importance of exercise as a non-pharmacological treatment option is emphasized, and it is aimed at making a significant contribution to the wide acceptance and application of such treatments.

ELIGIBILITY:
Inclusion Criteria:

* Having a score of 60 points or above on the menstrual symptoms scale
* Having a regular menstrual cycle (24-35 days)
* Not doing any exercise regularly
* Being between the ages of 18 and 25
* Nulliparity
* Being cooperative and oriented
* Volunteering to participate in the study

Exclusion Criteria:

* Having a medical history of chronic disease (cardiopulmonary, neurological, thyroid gland diseases)
* Having a history of regular exercise
* Engaging in regular sexual activity
* Having undergone gynecological surgical procedures
* Using hormonal contraceptive drugs or intrauterine devices
* Using a drug that causes dysmenorrhea
* Pelvic pathology, pelvic inflammatory diseases, endometriosis, etc. Having a disease that causes secondary dysmenorrhea
* Using antidepressant medication
* Having acute musculoskeletal system problems

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | At baseline, on the most painful 1 day of Cycle 1 (each cycle is 28 days), and on the most painful 1 day of Cycle 2 (each cycle is 28 days).
  Lower abdomen, leg and low back pain were evaluated with the Visual Analog Scale
Menstrual symptoms questionnaire | At baseline, on the most painful 1 day of Cycle 1 (each cycle is 28 days), and on the most painful 1 day of Cycle 2 (each cycle is 28 days).
  menstrual symptoms were evaluated with the Menstrual Symptoms Questionnaire
Pittsburgh Sleep Quality Index | At baseline, on the most painful 1 day of Cycle 1 (each cycle is 28 days), and on the most painful 1 day of Cycle 2 (each cycle is 28 days).
  sleep quality was evaluated with the Pittsburgh Sleep Quality Index
Health-Related Quality of Life Assessment (SF 36 Short Form) | At baseline, on the most painful 1 day of Cycle 1 (each cycle is 28 days), and on the most painful 1 day of Cycle 2 (each cycle is 28 days).
  Quality of life was evaluated with the Health-Related Quality of Life Assessment (SF 36 Short Form)
Functional and Emotional Dysmenorrhea Questionnaire | At baseline, on the most painful 1 day of Cycle 1 (each cycle is 28 days), and on the most painful 1 day of Cycle 2 (each cycle is 28 days).
  functional and emotional status was evaluated with the Functional and Emotional Dysmenorrhea Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moradpour, R., "Resistance training improves primary dysmenorrhea symptoms in young girls: A randomized controlled trial", Journal of Physical Activity and Hormones, 3(3): 35-48 (2019).
- [Background] Brown J, Brown S. Exercise for dysmenorrhoea. Cochrane Database Syst Rev. 2010 Feb 17;(2):CD004142. doi: 10.1002/14651858.CD004142.pub2. PMID 20166071
- [Background] Carroquino-Garcia P, Jimenez-Rejano JJ, Medrano-Sanchez E, de la Casa-Almeida M, Diaz-Mohedo E, Suarez-Serrano C. Therapeutic Exercise in the Treatment of Primary Dysmenorrhea: A Systematic Review and Meta-Analysis. Phys Ther. 2019 Oct 28;99(10):1371-1380. doi: 10.1093/ptj/pzz101. PMID 31665789
- [Background] Motahari-Tabari N, Shirvani MA, Alipour A. Comparison of the Effect of Stretching Exercises and Mefenamic Acid on the Reduction of Pain and Menstruation Characteristics in Primary Dysmenorrhea: A Randomized Clinical Trial. Oman Med J. 2017 Jan;32(1):47-53. doi: 10.5001/omj.2017.09. PMID 28042403